CLINICAL TRIAL: NCT04862221
Title: A Phase 2b, Double-Blind, Three Arm, Randomized, Placebo Controlled Trial With Restricted Response Adaptive Randomization Testing the Efficacy and Safety of High Dose Methylprednisolone or Equine Anti-Thymocyte Globulin as Treatment for Acute Liver Failure in Pediatric Patients
Brief Title: TReatment for ImmUne Mediated PathopHysiology
Acronym: TRIUMPH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PALF IRN/TRIUMPH; U01DK062436 (NIH)
Record Dates: First submitted 2021-04-23; First posted 2021-04-27 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Acute Liver Failure; Fulminant Hepatic Failure; Hepatic Encephalopathy; Acute Liver Injury; Immune Dysregulation
Keywords: hepatic insufficiency; liver diseases; liver failure; anti-thymocyte agents
MeSH Terms: conditions — Liver Failure, Acute; Hepatic Encephalopathy; Hepatic Insufficiency; Liver Diseases; Liver Failure | interventions — Methylprednisolone; Methylprednisolone Hemisuccinate; Antilymphocyte Serum; Prednisolone; Sodium Chloride; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- High-dose methylprednisolone (Experimental): Intravenous methylprednisolone at an initial dose of 10 mg/kg/day for 3 days, 5 mg/kg/day on day 4.
  Interventions: Drug: High-dose methylprednisolone; Drug: Prednisolone
- Equine anti-thymocyte globulin (Experimental): Intravenous equine anti-thymocyte globulin at a dose of 40 mg/kg/day for 4 days.
  Interventions: Drug: Equine anti-thymocyte globulin; Drug: Prednisolone; Drug: Diphenhydramine; Drug: Methylprednisolone
- Supportive care (Placebo Comparator): Supportive care will be administered as determined by the clinical team at participating clinical sites in accordance with their local practices and standards.
  Interventions: Drug: Placebo for prednisolone; Drug: Placebo for infusions

INTERVENTIONS:
Drug: High-dose methylprednisolone — Subjects in the high-dose methylprednisolone arm will receive an initial dose of methylprednisolone IV 10 mg/kg/day for 3 days and 5 mg/kg/day on Day 4. Normal saline will be used as placebo pre-medications and infusions given at the same volume and duration as the eATG infusions.
  Other Names: Solu-Medrol
  Arms: High-dose methylprednisolone
Drug: Equine anti-thymocyte globulin — Subjects will receive eATG IV 40 mg/kg/day on Days 1- 4. Day 1 eATG infusion is run over 8 hours and Day 2-4 infusions are run over 4 hours.
  Other Names: ATGAM
  Arms: Equine anti-thymocyte globulin
Drug: Prednisolone — Subjects will receive prednisolone 1 mg/kg on Days 5-13 followed by a gradual taper with discontinuation at 42 Days as indicated below.
  Days 5 - 13 Prednisolone PO 1 mg/kg/day (max 50 mg/day)
  Days 14- 20 Prednisolone PO 0.5 mg/kg/day (max 25 mg/day)
  Days 21 - 27 Prednisolone PO 0.3 mg/kg/day (max 15 mg/day)
  Days 28 - 34 Prednisolone PO 0.1 mg/kg/day (max 5 mg/day)
  Days 35 - 41 Prednisolone PO 0.1 mg/kg every OTHER day (max 5 mg every other day)
  Day 42 Discontinue
  Other Names: 15 mg/mL oral solution National Drug Code: 0121-0885-08
  Arms: Equine anti-thymocyte globulin; High-dose methylprednisolone
Drug: Placebo for prednisolone — Subjects will receive 1 mg/kg/day of oral placebo for prednisolone on days 5-13 followed by a gradual taper to discontinuation at 42 days as indicated below. Subjects receiving oral placebo will be given a solution that closely resembles the treatment drug.
  Days 5 - 13 Placebo for Prednisolone PO 1 mg/kg/day (max 50 mg/day)
  Days 14- 20 Placebo for Prednisolone PO 0.5 mg/kg/day (max 25 mg/day)
  Days 21 - 27 Placebo for Prednisolone PO 0.3 mg/kg/day (max 15 mg/day)
  Days 28 - 34 Placebo for Prednisolone PO 0.1 mg/kg/day (max 5 mg/day)
  Days 35 - 41 Placebo for Prednisolone PO 0.1 mg/kg every OTHER day (max 5 mg every other day)
  Day 42 Discontinue
  Arms: Supportive care
Drug: Placebo for infusions — Subjects randomized to the supportive care alone arm will receive normal saline in place of all study treatments (skin test, premedication and IV infusions) on Days 1-4 given at the same volume and duration as the eATG infusions.
  Other Names: 0.9% Sodium chloride
  Arms: Supportive care
Drug: Diphenhydramine — Subjects in the eATG arm will receive pre-treatment medication diphenhydramine IV 1 mg/kg prior to start of eATG infusion.
  Other Names: Benadryl
  Arms: Equine anti-thymocyte globulin
Drug: Methylprednisolone — Subjects in the eATG arm will receive pre-treatment medication methylprednisolone IV 1 mg/kg prior to start of eATG infusion.
  Other Names: Solu-Medrol
  Arms: Equine anti-thymocyte globulin

SUMMARY:
TReatment for ImmUne Mediated PathopHysiology (TRIUMPH) is a multi-center, three arm, randomized, controlled trial of immunosuppressive therapy for children with acute liver failure. The study will determine if suppressing inflammatory responses with either corticosteroids or equine anti-thymocyte globulin therapy improves survival for children with this rare, life-threatening condition.

DETAILED DESCRIPTION:
Pediatric Acute Liver Failure (PALF) is a rare, devastating condition that affects an estimated 250 children per year in North America, causing death in approximately 15% and the need for liver transplantation in an additional 20-30%. In the majority of cases, a specific cause of the liver injury is never determined. Recent research supports the theory that many of these patients have liver injury related to a hyperinflammatory immune response to everyday infections or environmental exposures. There is strong evidence to show that equine anti-thymocyte globulin and methylprednisolone slow the body's response to inflammation and improve the recovery of patients with other immune disorders and thus, may help patients with acute liver failure.

This is a phase 2b, double-blind, three arm, randomized, placebo controlled trial with restricted response adaptive randomization. The primary objective is to determine the efficacy and safety of high-dose methylprednisolone or equine anti-thymocyte globulin (eATG or ATGAM®) as compared to supportive care alone (placebo) for the treatment of acute liver failure in pediatric patients.

Approximately 160 patients who are equal to or greater than ≥ 1 and less than ≤ 18 years of age with pediatric acute liver failure (PALF) of undetermined etiology will be randomized to receive either high-dose methylprednisolone (Treatment 1) or eATG (ATGAM®) (Treatment 2) or supportive care alone (Treatment 3) on days 1 to 4 after study enrollment, followed by a gradual prednisolone taper (for the two active treatment arms 1 and 2) or a placebo taper (for treatment arm 3) on days 5 to 42.

The follow-up period includes visits at 1 week (Day 7), 2 weeks (Day 14), and 3 weeks (Day 21) after the day the participant started in the study. Early follow-up assessments will be performed either in the inpatient or ambulatory setting since some participants may be discharged before Day 7. In addition, families will be contacted by phone or email to schedule each follow-up at the study site for the 6 week, 3 month, 6 month and 12 month study visits.

This study will also include a prospective observational cohort study of up to 50 patients with PALF who meet the randomized controlled trial (RCT) eligibility criteria but who decline randomization in the RCT and are willing to provide longitudinal observational data.

The findings of this trial have the potential to shift the treatment paradigm in PALF and advance the basic understanding of immune dysregulation disorders in childhood. The network includes 20 of the largest and most active pediatric liver centers in the US who have organized to support rigorous testing of the efficacy and safety of immunosuppressive therapy for these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with liver injury of ≤ 6 weeks duration resulting in an international normalization ratio (INR) of ≥ 1.5 or < 2.0 (not corrected by vitamin K) with evidence of hepatic encephalopathy (HE), INR of ≥ 1.5 or < 2.0 for at least 7 days duration without evidence of HE or INR ≥ 2.0 without evidence of HE.
2. Age is greater than or equal to 1 year and less than 18 years of age.
3. Patient or their legally authorized representative(s) (LAR) must consent (and assent, if applicable) to be in the study and must have signed and dated an approved informed consent form which conforms to federal and institutional guidelines.
4. Females of reproductive potential should not plan on conceiving children during the study and must agree to use a medically accepted form of contraception.

Exclusion Criteria:

1. Evidence of active infection with Hepatitis A, B, C, E or evidence of acute herpes simplex virus (HSV) or adenovirus infection
2. Travel within the past 3 months to an area highly endemic for Hepatitis E
3. Diagnosis of hemophagocytic lymphohistiocytosis (HLH) Note: Patients with a history of consanguinity and/or central nervous system (CNS) dysfunction that is exaggerated compared to the degree of liver dysfunction (as judged by the site investigator) will not be enrolled until results of rapid genetic testing are available. Turn-around time for genetic testing results is estimated to be 72-96 hours.
4. Aplastic anemia as defined by standardized criteria [1] diagnosed prior to enrollment
5. Diagnosis of autoimmune Hepatitis (AIH)
6. Diagnosis of acute Wilson disease
7. Diagnosis of inborn error of metabolism Note: Suspicion of metabolic disease is not an exclusion for entry into the Trial.
8. Diagnosis of acute drug or toxin-induced liver injury
9. History of recreational drug use within the past 4 weeks
10. Therapy with an immunosuppressive agent, including chemotherapy, biological therapies or an experimental drug or device within the past 6 weeks
11. Liver injury due to ischemia
12. Liver dysfunction diagnosed more than 6 weeks prior to screening
13. History of allergy to horse dander
14. Sepsis
15. Imminent risk of death as judged by the clinical site investigator, including but not limited to; signs of cerebral herniation at the time of enrollment and presence of intractable arterial hypotension
16. Solid organ or stem cell transplant recipient
17. Pregnant or breast-feeding at the time of proposed study entry
18. Clinical AIDS or HIV positive
19. History of any form of malignant neoplasm and/or tumors treated within five years prior to study entry (other than non-melanoma skin cancer or in situ cervical cancer) or where there is current evidence of recurrent or metastatic disease
20. Received a live-virus vaccine within 4 weeks of study entry
21. Patients with positive respiratory secretion testing for respiratory viral infection including SARS-CoV-2, influenza and respiratory syncytial virus only if they also have declining respiratory function
22. Psychiatric or addictive disorders that would preclude obtaining informed consent/assent
23. Patient is unwilling or unable to adhere with study requirements and procedures
24. Currently receiving other experimental therapies

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 163 (Estimated)
Dates: Start 2022-02-09 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Survival with native liver (SNL) | 21 days
  Alive and without a liver transplant 21 days following randomization

SECONDARY OUTCOMES:
Survival with native liver (SNL) | 180 days
  Alive and without a liver transplant 6 months (180 days) following randomization

CONTACTS AND LOCATIONS:
Overall Officials: Estella M Alonso, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago; Valerie L Durkalski-Mauldin, PhD, Principal Investigator — Medical University of South Carolina; Ed Doo, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK); Averell Sherker, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (24):
- United States (24):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital, Palo Alto, California
  - Rady Children's Hospital, San Diego, California
  - University of California San Francisco Benioff Children's Hospital, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Yale New Haven Children's Hospital, New Haven, Connecticut
  - Children's Healthcare of Atlanta - Arthur M. Blank Hospital, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Children's Hospital Boston, Boston, Massachusetts
  - The Children's Mercy Hospital, Kansas City, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - The Mount Sinai Medical Center, New York, New York
  - NYP Morgan Stanley Children's Hospital, New York, New York
  - Duke University Medical Center - Duke Children's, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Children's, Cleveland, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Children's Hospital Vanderbilt, Nashville, Tennessee
  - UT Southwestern Medical Center Children's Health, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Data will be available at the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) Central Repository. The public use dataset, along with the study protocol, the data dictionary, annotated case report forms and a brief set of instructions ("Readme" file) will be provided.
Supporting Information: Study Protocol
Time Frame: Release of the public use dataset will follow the NIDDK guidelines that study data analyzed for publications must be shared with the broader scientific community at the time of publication. Also, the study data analyzed for publications will be submitted to the NIDDK-CR when the manuscript is accepted for publication or at the time of publication.
URL: https://repository.niddk.nih.gov/home/